CLINICAL TRIAL: NCT04813822
Title: A Phase 2, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Efficacy and Safety of Miconazole Nitrate 2% + Domiphen Bromide Vaginal Cream in the Treatment of Subjects With Acute Vulvovaginal Candidiasis
Brief Title: Study Evaluating the Efficacy and Safety of Miconazole Nitrate + Domiphen Bromide Vaginal Cream in the Treatment of Subjects With Acute Vulvovaginal Candidiasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aesculape CRO Belgium BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FHP-2021-2-26
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Acute Vulvovaginal Candidiasis
MeSH Terms: interventions — Miconazole; domiphen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Miconazole Nitrate 2% + Domiphen Bromide Low Dose Vaginal Cream (Experimental): The content of one applicator (5 g cream) is administered intravaginally once daily for 7 days.
  Interventions: Drug: Miconazole Nitrate 2% + Domiphen Bromide Low Dose
- Miconazole Nitrate 2% + Domiphen Bromide High Dose Vaginal Cream (Experimental): The content of one applicator (5 g cream) is administered intravaginally once daily for 7 days.
  Interventions: Drug: Miconazole Nitrate 2% + Domiphen Bromide High Dose
- Gyno-Daktarin® Vaginal Cream (Active Comparator): The content of one applicator (5 g cream) is administered intravaginally once daily for 7 days.
  Interventions: Drug: Miconazole Nitrate 2%

INTERVENTIONS:
Drug: Miconazole Nitrate 2% + Domiphen Bromide Low Dose — Dosage 1
  Arms: Miconazole Nitrate 2% + Domiphen Bromide Low Dose Vaginal Cream
Drug: Miconazole Nitrate 2% + Domiphen Bromide High Dose — Dosage 2
  Arms: Miconazole Nitrate 2% + Domiphen Bromide High Dose Vaginal Cream
Drug: Miconazole Nitrate 2% — Active Comparator
  Arms: Gyno-Daktarin® Vaginal Cream

SUMMARY:
This study is a multicentre, three-arm, double-blind, randomized controlled, parallel-group, comparative phase II clinical trial to evaluate miconazole nitrate 2% + domiphen bromide vaginal cream in subjects with acute vulvovaginal candidiasis.

DETAILED DESCRIPTION:
Females aged 18-50 years with a clinical diagnosis of an acute VVC episode at Screening Visit will be randomly assigned to either miconazole nitrate 2% + low or high dose of domiphen bromide vaginal cream or to the comparator product Gyno-Daktarin® vaginal cream (miconazole nitrate 2%). The creams will be applied for 7 days and subjects will be followed up for 12 weeks.

ELIGIBILITY:
Main inclusion criteria:

1. Subjects must be generally healthy, non-pregnant females, 18-50 years of age at Screening Visit.
2. Subjects must have an acute VVC episode at Screening Visit, defined as a total signs and symptoms score of ≥3 and a positive KOH wet mount preparation or Gram stain from a vaginal smear revealing filamentous hyphae/pseudohyphae and/or budding yeast cells.

Main exclusion criteria :

1. Subjects with the presence of concomitant vulvovaginitis caused by other pathogens at Screening Visit, or any other infection that requires antibiotic treatment.
2. Subjects with visible condylomas on vulvovaginal examination at Screening Visit.
3. Subjects with the presence or a history of another vaginal or vulvar condition(s) that in the Investigator's opinion would confound the interpretation of the clinical response.
4. Subjects with a history of cervical cancer.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with clinical cure | First follow-up visit (Day 15)
  Resolution of the VVC signs and symptoms that were present at Screening Visit (Baseline)
The proportion of subjects with mycological eradication | First follow-up visit (Day 15)
  A culture negative vaginal swab for growth of baseline Candida species
The proportion of subjects with overall therapeutic success | First follow-up visit (Day 15)
  Achievement of both clinical cure and mycological eradication

SECONDARY OUTCOMES:
The proportion of subjects with clinical cure | First follow-up visit through Week 12
  Resolution of the VVC signs and symptoms that were present at Screening Visit (Baseline)
The proportion of subjects with mycological eradication | First follow-up visit through Week 12
  A culture negative vaginal swab for growth of baseline Candida species at Day 15, a culture and PCR negative vaginal swab for growth of baseline Candida species on the Other follow-up visits
The proportion of subjects with overall therapeutic success | First follow-up visit through Week 12
  Achievement of both clinical cure and mycological eradication
Change from Baseline in vulvovaginitis symptom questionnaire total score | Through Week 12
  VSQ: Vulvovaginal symptoms questionnaire
Change from Baseline in the EQ-5D questionnaire total score | Through Week 12
  EQ-5D: health-related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Deslypere, MD, Study Director — Aesculape CRO Belgium BV
Locations (6):
- Belgium (6):
  - UZ Antwerpen - Gynaecology department, Edegem, Antwerpen
  - Femicare vzw, Tienen, Brabant
  - Fertiliteitscentrum Dr. Decleer Aalter, Aalter, East Flanders
  - UZ Gent - Gynaecology department, Ghent, East Flanders
  - Dr. Goessens - Dr. Houben, Private practice - Gynaecology, Bruges, West Flanders
  - Dr. Philip Loquet, Private practice - Gynaecology, Antwerp